CLINICAL TRIAL: NCT01471379
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy of Milnacipran in the Treatment of Irritable Bowel Syndrome
Brief Title: Milnacipran (Savella) in Irritable Bowel Syndrome (IBS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to recruitment difficulties the study is terminated.
Sponsor: Spencer Dorn, MD, MPH (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Spencer Dorn, MD, MPH, Assistant Professor of Medicine, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-1105a
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; IBS; Savella; Milnacipran; Abdominal Pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (50mg - 100mg) (Experimental): Group A will begin treatment with Milnacipran 50mg BID (n=20) during Phase I and will be increased to 100mg BID during Phase II
  Interventions: Drug: Milnacipran
- Group B (50mg x12) (Active Comparator): Subjects in this arm will be maintained at Milnacipran 50mg BID for the entirety of the 12 weeks of the study.
  Interventions: Drug: Milnacipran
- Group C (Placebo - 50mg) (Placebo Comparator): Group C will begin treatment with Placebo BID (n=20) during Phase I and will be given 50mg BID during Phase II
  Interventions: Drug: Milnacipran; Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — 50mg Milnacipran PO, BID, for 6 weeks.
  Other Names: Savella
  Arms: Group A (50mg - 100mg); Group C (Placebo - 50mg)
Drug: Milnacipran — Milnacipran, 100mg PO, BID, for six weeks
  Other Names: Savella
  Arms: Group A (50mg - 100mg)
Drug: Milnacipran — Milnacipran, 50mg PO BID for 12 weeks
  Other Names: Savella
  Arms: Group B (50mg x12)
Drug: Placebo — Inactive pill, identical in shape, size, and appearance to active drug, PO, BID.
  Arms: Group C (Placebo - 50mg)

SUMMARY:
Purpose: The investigators are proposing to examine the use of Savella® (Milnacipran) for treating irritable bowel syndrome (IBS) in women.

Participants: Eligible participants will meet the Rome III diagnostic criteria for IBS.

Procedures: This study will observe patients treated with Savella® as well as patients treated with a placebo (pill with no active drug). The investigators will monitor and compare several patient and symptom related outcomes, as well as evaluate health related quality of life, psychological distress and related psychosocial measures to determine if the addition of Savella® improves clinical pain response as well as secondary outcomes including quality of life.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common functional gastrointestinal disorder characterized primarily by abdominal pain associated with bowel dysfunction. Like many other painful functional somatic syndromes (e.g. fibromyalgia) the pathophysiology of IBS includes abnormal responses to pain and dysregulation of brain-body pain pathways. IBS affects up to 10% of the population, is a leading reason for visits to gastroenterologists and primary care doctors, and, in the United States, annually accrues health care costs over $20 billion.

In their practice the investigators use centrally acting agents to treat IBS. Historically, the investigators have used tricyclic antidepressants based on results of clinical trials, including our NIH funded trial on desipramine. Nonetheless, these agents can produce side effects that limit their full application. More recently the investigators have begun to use SNRIs because they have been shown to benefit for various pain syndromes like diabetic neuropathy, fibromyalgia. The initial impression is that Milnacipran helps improve IBS symptoms and global well being. There is now a need to systematically determine Milnacipran's value for IBS.

ELIGIBILITY:
Inclusion Criteria:

* Meet Rome III criteria for IBS and have no red flags.
* Must have had a colonoscopy within the previous 5 years to exclude inflammatory or other bowel disease
* Be fluent and literate in English
* Must either be of non-childbearing potential or agree to utilize approved birth control for the duration of the study

Exclusion Criteria:

* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the GI tract within 6 months prior to screening, or active disease within 6 months prior to screening.
* Any other diagnosis to explain the abdominal pain,
* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, neurologic, psychiatric or any disease that may interfere with the subject successfully completing the trial
* Hepatic dysfunction (ALT [SGPT] or AST [SGOT] >3 times the upper limit of normal) or renal impairment (serum creatinine > 2mg/dL)
* Has disease affecting electrolytes balance, such as SIADH with serum Sodium less than 130mmol/L
* Any evidence of or treatment of malignancy (other than localized basal cell, squamous cell skin cancer or cancer in situ that has been resected) within the previous year
* Any surgery on the stomach, small intestine or colon, excluding appendectomy
* A major psychiatric disorder (DSM-III-R or DSM-IV) including major depression or other psychoses that has required hospitalization in the last 1 year.
* History of attempted suicide or uncontrolled bipolar disorder.
* Currently using antidepressants for psychiatric conditions like major depression. Use of TCA or SSRI class antidepressant acceptable if being used specifically for treatment of bowel symptoms and patient is willing to taper off the medication
* Previous use of Milnacipran or other SNRI antidepressant (duloxetine, venlafaxine, desvenlafaxine)
* A diagnosis of seizure disorder
* A diagnosis of glaucoma
* Currently taking heparin or warfarin

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spencer D Dorn, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Center for Functional GI and Motility Disorders, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited from community using University of North Carolina (UNC) mass email system, newspaper advertisement and UNC gastrointestinal (GI) clinic referral.
Pre-assignment Details: Subjects undergo screening labs and questionnaires to make sure subjects are healthy and don't have any underlying conditions. Subjects who had clinically significant labs or Hospital Anxiety and depression scale(HADS)score more than 17 were excluded.
Groups:
- Group A (50mg - 100mg): Group A will begin treatment with Milnacipran 50mg twice a day (BID) (n=20) during Phase I and will be increased to 100mg BID during Phase II
  Milnacipran : 50mg Milnacipran per orally (PO), BID, for 6 weeks.
  Milnacipran : Milnacipran, 100mg PO, BID, for six weeks
- Group B (50mg x12): Subjects in this arm will be maintained at Milnacipran 50mg BID for the entirety of the 12 weeks of the study.
  Milnacipran : Milnacipran, 50mg PO BID for 12 weeks
- Group C (Placebo - 50mg): Group C will begin treatment with Placebo BID (n=20) during Phase I and will be given 50mg BID during Phase II
  Milnacipran : 50mg Milnacipran PO, BID, for 6 weeks.
  Placebo : Inactive pill, identical in shape, size, and appearance to active drug, PO, BID.
Period: Overall Study
Arm/Group | Group A (50mg - 100mg) | Group B (50mg x12) | Group C (Placebo - 50mg)
Started | 1 | 1 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Study terminated | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated early resulting in a small number of subjects enrolled leaving the ability to analyze only certain categories.
Groups:
- Group A (50mg - 100mg): Group A will begin treatment with Milnacipran 50mg BID (n=20) during Phase I and will be increased to 100mg BID during Phase II
  Milnacipran : 50mg Milnacipran PO, BID, for 6 weeks.
  Milnacipran : Milnacipran, 100mg PO, BID, for six weeks
- Total: Total of all reporting groups
Arm/Group | Group A (50mg - 100mg) | Group B (50mg x12) | Group C (Placebo - 50mg) | Total
Number analyzed (Participants) | 1 | 1 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 1 | 1 |  | 2
  >=65 years | 0 | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (0) | 66 (0) |  | 56.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 |  | 2
  Male | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pain Response
Description: Visual Analog Scale (VAS) scores (range 0-100 mm; 0 = none, 100 = worst pain) were recorded for pain before the beginning of the study, at 6 weeks of treatment and at the end visit i.e. 10 weeks. Ideally, VAS would have been administered at the 12th week; however, subject was terminated at the 10th week visit. A positive pain response (ie pain relief) was defined as >30% decrease in the VAS score between baseline and the final study visit.
Time Frame: Twelve Weeks
Measure: Number; unit: participants
Groups:
- Group A (50mg - 100mg): Group A begins treatment with Milnacipran 50mg BID (n=20) during Phase I and will be increased to 100mg BID during Phase II
  Milnacipran : 50mg Milnacipran PO, BID, for 6 weeks.
  Milnacipran : Milnacipran, 100mg PO, BID, for six weeks
Arm/Group | Group A (50mg - 100mg) | Group B (50mg x12) | Group C (Placebo - 50mg)
Number analyzed (Participants) | 1 | 0 | 0
participants | 0 |  |

2. Secondary Outcome: Quality of Life ( IBS-QOL)
Description: After six weeks of treatment with Milnacipran, treatment groups were compared with placebo for clinically significant improvement in IBS-QOL. 11 point reduction in IBS-QOL compared to baseline was considered as clinically significant improvement.
Time Frame: Six Weeks
Arm/Group | Group A (50mg - 100mg) | Group B (50mg x12) | Group C (Placebo - 50mg)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Subject Self Reported Adequate Relief of Pain
Description: The study sought to determine if the Milnacipran arms had a greater proportion of adequate relief over the placebo group. Subjects were asked to answer 'yes' or 'no' as to whether or not they had adequate relief of pain due to irritable bowel syndrome.
Time Frame: Twelve Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Group A (50mg - 100mg) | Group B (50mg x12) | Group C (Placebo - 50mg)
Number analyzed (Participants) | 1 | 0 | 0
percentage of participants | 0 |  |

4. Secondary Outcome: Treatment Efficacy Questionnaire (TEQ)
Description: Treatment Efficacy Questionnaire is a measure of treatment effectiveness. The score ranges from 1 to 48, 1 is minimum score and 48 is the maximum score. The investigators was looking to see if the Milnacipran treatment groups have a higher proportion of subjects with significant improvement in efficacy, judged as a TEQ score of >28, compared to placebo group.
Time Frame: Twelve Weeks
Population: Only one subject was enrolled and was analyzed even though subject did not complete the study.
Measure: Number; unit: percentage of subject with score >28
Arm/Group | Group A (50mg - 100mg) | Group B (50mg x12) | Group C (Placebo - 50mg)
Number analyzed (Participants) | 1 | 0 | 0
percentage of subject with score >28 | 0 |  |

5. Secondary Outcome: Dose Related Incremental Benefit in Pain Reduction Based on VAS
Description: The investigator was looking to see if, for group A, when increased from 50 mg BID to 100 mg BID there is significant improvement of pain scores i.e. 30% pain reduction, and for group C, if there was significant improvement of pain scores when switched from placebo to 50 mg BID of Milnacipran
Time Frame: 12 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Group A (50mg - 100mg) | Group B (50mg x12) | Group C (Placebo - 50mg)
Number analyzed (Participants) | 1 | 0 | 0
percentage of participants | 0 |  |

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Group A (50mg - 100mg) | Group B (50mg x12) | Group C (Placebo - 50mg)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (50mg - 100mg) (N=1) | Group B (50mg x12) (N=0) | Group C (Placebo - 50mg) (N=0)
hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No